CLINICAL TRIAL: NCT04424186
Title: Effect of Measuring Vital Signs and Coherent Rehabilitation in Primary and Secondary Sectors in Older Adults After Hip Fracture Surgery
Brief Title: 'Rehabilitation for Life'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kolding Sygehus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: SLB-Phys-06-2020
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hip Fractures
Keywords: Rehabilitation; cross-sectorial cooperation; older
MeSH Terms: conditions — Hip Fractures | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: A cluster-randomized stepped wedge study. A design that is initiated with a period without interventions followed by a form of cross-over, in which each cluster systematic cross from control to intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Rehabilitation for Life' (Experimental): Vital sign measurement and rehabilitation
  Interventions: Other: 'Rehabilitation for Life'
- Usual care and rehabilitation (Active Comparator): Usual care and rehabilitation provided in primary and secondary sectors
  Interventions: Other: Usual care and rehabilitation

INTERVENTIONS:
Other: 'Rehabilitation for Life' — An empowerment-oriented cross-sectorial program including vital sign measurement and systematic progressive rehabilitation combined with convenient access for collaboration among professionals.
  Arms: 'Rehabilitation for Life'
Other: Usual care and rehabilitation — The care and rehabilitation usual provided to patients after hip fracture surgery
  Arms: Usual care and rehabilitation

SUMMARY:
Despite implementing hospital quality programs after hip fracture surgery older adults often experience a decline in the level of physical function, reduced quality of life; and the mortality and readmission rates are high.

Early mobilization is important in order to prevent loss of muscle mass; however to prevent morbidity an early start of strength training is also necessary. Furthermore, the risk of complications, morbidity, and mortality are associated with insufficient management of pain.

The project aims to examine the effect of measuring vital signs and consistent rehabilitation in the primary and secondary sectors in older adults after hip fracture surgery.

Method/ design:

The study is a cluster-randomized stepped wedge study. Participants will be recruited among patients admitted to an orthogeriatric ward who are 65 years of age or older and citizens in one of six municipalities. Participants are also the health professionals in the orthogeriatric ward and the six municipalities.

The six municipalities form six clusters, which are randomized, and every three-month one cluster cross from control to intervention.

The study compares usual practice (control) to an intervention named 'Rehabilitation of Life'. An intervention best described as an empowerment-oriented cross-sectorial program including vital sign measurement and systematic progressive rehabilitation and combined with convenient access for collaboration among professionals.

Primary outcomes: Timed Up and Go (TUG) measured 2 months after the time of operation.

The investigators hypothesize that 'Rehabilitation of Life' for older adults with a hip fracture will result in a significant reduced TUG-score in comparison to a practice not offering 'Rehabilitation of Life'.

And as the study is organised across two sectors, the Cumulated Ambulation Score (CAS) makes a second primary outcome. It is hypothesised that patients in the intervention group will achieve a significantly reduced TUG score compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a hip fracture
* Patients of 65 years of age or older
* Patients admitted to an orthogeriatric ward
* Patient who are citizens in one og three municipalities

Exclusion Criteria:

* Patients discharged for permanent residence in nursing homes
* Patients who cannot participate in a conversation
* Terminal registered patients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 339 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Timed up and go | Two months after the time of operation
  Measures functional mobility, as the time in seconds it takes a person to rise from a chair with arms, walk 3 m and return to the chair. A higher scores mean a worse outcome
Cumulated Ambulation Score (CAS) | One months after the time of operation
  Measures basic mobility. The score 0-6. Higher scores mean a better outcome

SECONDARY OUTCOMES:
Timed up and go | Three and six months after the time of operation
  Measures functional mobility, as the time in seconds it takes a person to rise from a chair with arms, walk 3 m and return to the chair. A higher scores mean a worse outcome
Barthel-20 | 2, 3, 6 and 12 months after the time of surgery
  A validated tool used to assess the patient's need for help to perform acitivities of daily living

OTHER OUTCOMES:
Eq-5D | 2, 3, 6 and 12 months after the time of surgery
  A standardised questionnaire used to assess the patients health-related quality of life and function
Mortality 30 days and 1 year. | Mortality measured after 30 days and one year
  Mortality
Readmission | Readmission measured 30 days after discharge
  Readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: Inge Bruun, post doc, Study Chair — The Region of Southern Denmark and University of Southern Denmark
Locations (1):
- Inge Bruun, Kolding, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ipsen JA, Pedersen LT, Viberg B, Norgaard B, Suetta C, Bruun IH. Rehabilitation for life: the effect on physical function of rehabilitation and care in older adults after hip fracture-study protocol for a cluster-randomised stepped-wedge trial. Trials. 2022 May 7;23(1):375. doi: 10.1186/s13063-022-06321-w. PMID 35526010